CLINICAL TRIAL: NCT01021761
Title: A Comparison of Prostaglandin E2 (PGE2) Inhibition of Acuvail, Xibrom and Nevanac in Patients Undergoing Phacoemulsification
Brief Title: A Comparison of Prostaglandin E2 (PGE2) Inhibition of Acuvail(Ketorolac 0.45%), Xibrom (Bromfenac 0.09%)and Nevanac (Nepafenac)in Patients Undergoing Phacoemulsification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frank A. Bucci, Jr., M.D. (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Frank A. Bucci, Jr., M.D., Medical Director, Bucci Laser Vision Institute
Organization: Bucci Laser Vision Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009 0199
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — Ketorolac Tromethamine; Ketorolac; bromfenac; nepafenac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Xibrom (Active Comparator): Xibrom to be given 1 drop 2 times (BID) the day before surgery and 3 doses pre op the day of surgery prior to surgery
  Interventions: Drug: Bromfenac
- Nevanac (Active Comparator): Nevanac to be given 1 drop 2 times (BID) the day before surgery and 3 doses pre op the day of surgery prior to surgery
  Interventions: Drug: nepafenac
- Acuvail (Active Comparator): Acuvail to be given preoperatively. One drop 2 times (BID), 1 day pre op and day of surgery 3 doses prior to surgery.
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — ketorolac to be given 1 drop BID the day before surgery and 3 doses pre op the day of surgery prior to surgery
  Other Names: Acuvail
  Arms: Acuvail
Drug: Bromfenac — Drug to be given 1 drop BID the day before surgery and 3 doses pre op the day of surgery prior to surgery
  Other Names: Xibrom
  Arms: Xibrom
Drug: nepafenac — drug to be given 1 drop BID the day before surgery and 3 doses pre op the day of surgery prior to surgery
  Other Names: Nevanac
  Arms: Nevanac

SUMMARY:
Approximately 126 subjects scheduled to undergo cataract surgery by phacoemulsification, will be randomized in an even allocation (1:1:1) to either Acuvail, Xibrom or Nevanac. Subjects will be instructed to begin dosing the study medication in the operative eye the day before surgery and continue dosing on the day of surgery. Beginning one hour before surgery 1 drop of study medication will be instilled by operating room staff approximately every 15 minutes for a total of 3 doses. At the designated time a paracentesis will be performed at the start of the cataract procedure and at least 0.15cc of aqueous humor will be collected. The sample will be immediately stored on dry ice and shipped to a laboratory for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older
* Scheduled for cataract surgery by phacoemulsification
* Subjects must be willing to comply with all study requirements and be willing to give informed consent

Exclusion Criteria:

* Any subject that has a history of uveitis or active iritis
* Subject can have o previous eye surgery with the exception of refractive surgery but not within 6 month
* No ocular use of prostaglandins within 2 weeks of surgery
* Use of oral, injectable or topical ophthalmic steroids, NSAIDs of immunosuppressants within 14 days prior to surgery
* Contraindications to nonsteroidal anti-inflammatory drugs (NSAIDs)
* Active ocular infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Bucci, Jr., MD, Principal Investigator — Bucci Laser Vision

RESULTS

PARTICIPANT FLOW:
Groups:
- Xibrom: Xibrom to be given 1 drop BID the day before surgery and 3 doses pre op the day of surgery prior to surgery
- Nevanac: Nevanac to be given 1 drop BID the day before surgery and 3 doses pre op the day of surgery prior to surgery
- Acuvail: Acuvail to be given preoperatively. One drop BID, 1 day pre op and day of surgery 3 doses prior to surgery.
Period: Overall Study
Arm/Group | Xibrom | Nevanac | Acuvail
Started | 42 | 42 | 42
Completed | 41 | 38 | 42
Not Completed | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xibrom | Nevanac | Acuvail | Total
Number analyzed (Participants) | 42 | 42 | 42 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 15 | 21 | 54
  >=65 years | 24 | 27 | 21 | 72
Age Continuous [Mean (Standard Deviation); unit: years] | 72 (31) | 74 (29) | 75 (30) | 74 (29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 26 | 81
  Male | 16 | 13 | 16 | 45
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 42 | 126

OUTCOME MEASURES:

1. Primary Outcome: Aqueous PGE2 Inhibition
Description: A spectroscopic quantification of PGE2 was performed on the aqueous humor samples collected with the results measured in pg/ml. PGE2 levels below 50 pg/ml were considered below the level of detection.
Time Frame: Day 4 of treatment
Population: Protocol specified 126 subjects to be enrolled and analysis was performed per protocol.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Xibrom | Nevanac | Acuvail
Number analyzed (Participants) | 42 | 42 | 42
pg/ml | 288.7 (226.05) | 320.4 (205.6) | 224.8 (164.87)

ADVERSE EVENTS:
Arm/Group | Xibrom | Nevanac | Acuvail
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes